CLINICAL TRIAL: NCT05666323
Title: Increasing Treatment for Obesity Among Underserved Populations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Ben B & Iris Margolis Private Foundation for Medical Research (Unknown)
Responsible Party: Principal Investigator, David Wetter, Director, University of Utah
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: HCI139694
Record Dates: First submitted 2022-12-16; First posted 2022-12-27 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — TM 1; Patient Navigation

STUDY DESIGN:
Intervention Model Description: This study will use a Sequential Multiple Assignment Randomized Trial (SMART) Design, which will allow investigators to address questions like those of traditional factorial design and assess dynamic treatment regimens to inform the development of adaptive interventions. An adaptive intervention contains a sequence of individually tailored decision rules that specify the intensity or type of intervention at critical points in the delivery of care. Modifying intensity or type of intervention over time can improve outcomes if an individual is not responding, or may reduce costs and patient burden if more resource intensive treatment is not necessary. As such, the proposed SMART design informs the development of adaptive and stepped care interventions, and the reduction in patient burden is particularly important to ensure that the interventions are as patient centered as possible.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Phase 1: TM1 (Experimental): Patients in the TM1 condition will be randomized to receive either an autonomy supportive message, or a directive motivational message.
  Interventions: Behavioral: Single Text Messaging (TM1)
- Phase 1: TM+ (Experimental): Patients in the TM+ condition will be randomized to receive 5 text messages in scheduled succession. These messages will be either an autonomy supportive message, or a directive motivational message.
  Interventions: Behavioral: Multiple Text Messaging (TM+)
- Phase 2: TM1 and PN (Experimental): Patients in the TM1 and PN condition will be randomized to receive either an autonomy supportive message, or a directive motivational message. Additionally, they will receive the option to talk with a Patient Navigator to receive MAPS coaching
  Interventions: Behavioral: Single Text Messaging (TM1); Behavioral: Patient Navigation (PN)
- Phase 2: TM1 continued (Experimental): Patients in the TM1 continued arm have the continued option to reply to the first text message in "Phase 1: TM1." They do not receive any additional intervention.
  Interventions: Behavioral: Single Text Messaging (TM1)
- Phase 2: TM+ and PN (Experimental): Patients in the TM+ and PN condition will be randomized to receive 3 additional either autonomy supportive messages, or directive motivational messages. Additionally, they will receive the option to talk with a Patient Navigator to receive MAPS coaching
  Interventions: Behavioral: Patient Navigation (PN); Behavioral: Multiple Text Messaging (TM+)
- Phase 2: TM+ continued (Experimental): Patients in TM+ continued will receive 3 additional either autonomy supportive messages, or directive motivational messages.
  Interventions: Behavioral: Multiple Text Messaging (TM+)

INTERVENTIONS:
Behavioral: Single Text Messaging (TM1) — Receives single text message
  Arms: Phase 1: TM1; Phase 2: TM1 and PN; Phase 2: TM1 continued
Behavioral: Patient Navigation (PN) — Receive phone calls from trained MAPS counselors
  Arms: Phase 2: TM+ and PN; Phase 2: TM1 and PN
Behavioral: Multiple Text Messaging (TM+) — Receives multiple scheduled text messages
  Arms: Phase 1: TM+; Phase 2: TM+ and PN; Phase 2: TM+ continued

SUMMARY:
The objective of this project is to evaluate strategies to increase patient engagement in evidence-based interventions (EBIs) for obesity. The scientific premise of the proposed project is based on: 1) substantial evidence that EBIs for obesity are effective but grossly underutilized, 2) promising results indicating that technology-based approaches such as text messaging may increase the reach of EBIs among underserved populations, 3) data demonstrating that repeated offers of treatment can substantially increase enrollment even among patients who are initially unmotivated, and 4) prior research highlighting the effectiveness of Motivation And Problem Solving (MAPS), a proactive coaching approach used to address barriers to improve patient enrollment in EBIs.

Thus, the proposed project will develop, implement, and evaluate two strategies for increasing the assessment and enrollment of University of Utah Medicaid patients in online EBIs for obesity: 1) Repeated offers of EBIs for obesity using text messaging and state of the science health communication strategies, 2) MAPS navigation/counseling among patients who do not enroll in EBIs in response to text messaging. The proposed project will provide critical data regarding the implementation of pragmatic and scalable interventions that are designed to increase the reach of existing EBIs for obesity among underserved populations. Most importantly, the project results lay the foundation for the widespread dissemination of strategies to increase use of EBIs for obesity across Utah, the Mountain West region, and the nation.

Project deliverables include 1) a text messaging intervention for facilitating connection to EBIs for obesity; 2) MAPS intervention for facilitating connection to EBIs for obesity; 3) implementation, adaptation, and optimization of these interventions for University of Utah Medicaid patients, 4) preliminary evidence for the efficacy of these two interventions in improving the reach of EBIs for obesity, and 5) creation of a plan for further dissemination.

DETAILED DESCRIPTION:
This study will use a Sequential Multiple Assignment Randomized Trial (SMART) Design, which will allow participants to address questions like those of traditional factorial design and assess dynamic treatment regimens to inform the development of adaptive interventions. An adaptive intervention contains a sequence of individually tailored decision rules that specify the intensity or type of intervention at critical points in the delivery of care. Modifying intensity or type of intervention over time can improve outcomes if an individual is not responding, or may reduce costs and patient burden if more resource intensive treatment is not necessary. As such, the proposed SMART design informs the development of adaptive and stepped care interventions, and the reduction in patient burden is particularly important to ensure that the interventions are as patient centered as possible.

The first randomization is a patient-level randomization to text messaging (single) versus text messaging (multiple) among eligible patients. The second randomization is a patient-level randomization to Motivation And Problem Solving (MAPS) coaching vs. no MAPS among the remaining patients in the text message conditions who do not enroll in the EBI. The primary outcome for this study is enrollment in an online EBI for obesity. IncentaHEALTH provides EBIs for obesity to the University of Utah Health system, either the Diabetes Prevention Program or Lifestyle Change Program. Their online Diabetes Prevention Program (DPP) is fully recognized by CDC.

Study Design:

To identify the cohort for the intervention, patient data will be extracted from the University of Utah EHR. Data fields will include variables such as age, gender, body mass index, pregnancy status, medical codes (e.g., ICD-10 for Type 1 and Type 2 diabetes), patient demographics (e.g., zip code, insurance status, preferred language, race/ethnicity); as well as contact information for text messaging and patient navigation. Patients who fit within the inclusion/exclusion criteria will be randomly selected and assigned to the conditions described below.

This study will take place in two Stages spanning a 6-12 month period. In Stage 1 (0 - 12 weeks), participants will be randomized to one of two conditions: Text Messaging 1 (Single text; hereafter referred to as TM1), or Text Messaging Plus (Multiple texts; hereafter referred to as TM+). The study team will use a 1:1 randomization ratio (TM1: TM+).

Prior to being contacted via text message, participants in the TM1 and TM+ conditions will receive an e-mail informing participants that they will be receiving communications from The University of Utah Health about the availability of a healthy lifestyle program. The e-mail will provide patients with information about how they can opt-out if they do not wish to receive these communications. Patients who do not have a valid e-mail address on file will be contacted via mail with instructions regarding how to opt-out.

Patients in the TM1 condition will receive one HIPAA-compliant bidirectional text message with the option to reply "yes" or opt out. The text will include a brief motivational message including information about DPP eligibility and the opportunity to enroll. Patients who reply "yes" will be contacted by IncentaHEALTH to enroll in the DPP or a similar lifestyle change program, depending on patient eligibility. Patients who enroll or opt out of receiving text messages will not be contacted again.

Patients in the TM+ condition will receive a HIPAA-compliant bidirectional text message weekly for the first 2 weeks and then every three weeks through week 12. Patients will receive text messages until they opt-out or reply "yes" to enroll. The text will include a brief motivational message including information about DPP eligibility and opportunity to enroll. Patients who reply "yes" will be contacted by IncentaHEALTH to enroll in the DPP or a similar lifestyle change program, depending on patient eligibility. Patients who enroll or opt out of receiving text messages will not be contacted again.

In Stage 2 of the study (weeks 13-24), patients will be randomized as follows:

Patients randomized to the TM1 condition in Stage 1 who did not respond to the single text message by 12 weeks (i.e., enroll in the EBI or opt out) will either be randomized to receive Motivational And Problem Solving (MAPS) counseling (TM1 & MAPS), or will not be contacted again (TM1 cont'd). Participants randomized to TM1 & MAPS will receive two MAPS calls during Stage 2.

Patients randomized to the TM+ condition in Stage 1 who did not respond to the text messages by 12 weeks (i.e., enroll in the EBI or opt out) will be randomized either to receive continued (monthly) text messages and MAPS counseling (TM+ & MAPS) or continued (monthly) text messages only (TM+ cont'd). Participants randomized to TM+ & MAPS will receive two MAPS calls during Stage 2.

Prior to being contacted by the MAPS counselors, participants randomized to the MAPS conditions in Stage 2 will receive one text message informing the participants that a MAPS counselor will call the participant about enrolling in a lifestyle change program. This text message will also provide participants with an opportunity to opt out from having a MAPS counselor call the participants.

Text Messaging Intervention

The study team will send bidirectional texts to patients. Text messages have been designed by the research team in consultation with the current research literature. All text messages will be sent using U Health's HIPAA compliant text messaging service, which has previously been utilized by our team. The text messaging service will retrieve the patient cohort from the study database to send the TMs to the patients. Every text message will include the option to opt out to cease receiving text messages at any time. Patients are routinely contacted by clinics via phone calls, emails, and text messages; therefore the text messages are not beyond the scope of routine care and correspondence.

Text messages will include a motivational message, the Diabetes Prevention Program phone number, and a simple two-touch response that directly connects interested patients to the Diabetes Prevention Program. Patients in the TM+ condition will be randomized to one of three types of motivational messages: 1) autonomy supportive motivational messaging; 2) directive motivational messaging; and 3) a combination of autonomy supportive and motivational messaging. Patients in the TM1 condition will be randomized to receive either an autonomy supportive message, or a directive motivational message. The two types of messages do not fundamentally alter the intervention and this will support exploratory analyses only.

Motivation And Problem Solving (MAPS) Intervention

MAPS is an empirically validated proactive coaching approach used to address barriers and motivate participants to engage in EBIs. Trained MAPS counselors will directly contact patients via secure telephone line to assess their motivation and provide counseling related to enrolling in the EBI. As with the text messages, patients can opt out of MAPS counseling at any time. University of Utah Health currently employs patient navigators and community health workers to perform patient navigation for various reasons (e.g., coordination of care, resource referral); therefore, patient navigation is not beyond the standard of care for patients.

IncentaHEALTH EBIs for obesity

IncentaHEALTH will triage interested patients into either online DPP or lifestyle change using a CDC risk assessment tool. Their lifestyle change program uses the same general components as the DPP. Both programs are designed to increase intake of fruits, vegetables, lean protein, and complex carbohydrates while monitoring portion size. Physical activity recommendations include cardiovascular and strength training, with a goal of approximately 30 minutes 5-6 days/week. Both are offered in English and Spanish, based on social cognitive theory, and provide personalized health coaching. Both include a website, Bluetooth wireless scale for weight monitoring, daily email/text message support, video exercise plans, customized meal plans, grocery lists, and incorporate skill building, social accountability, and reinforcement. Participants have unlimited online access to Health Coaches, who have at least a Bachelor's degree and certifications in personal training, nutrition, or wellness.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be adults aged 18+
* have a BMI of 30 or higher
* have had a primary care appointment within University of Utah Health within the past year
* speak English or Spanish as their primary language
* have a current Utah address
* are insured through Medicaid (University of Utah Health Plans).

Exclusion Criteria:

* patients may not have a diagnosis of Type 1 or Type 2 Diabetes
* being currently pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2022-03-23 (Actual); Primary Completion 2023-02-08 (Actual); Study Completion 2023-02-08 (Actual)

PRIMARY OUTCOMES:
Proportion of participants who were eligible, contacted, and enrolled in the trial. | at 12 weeks
  Proportion of participants who were eligible, contacted, and enrolled in the trial.

SECONDARY OUTCOMES:
Evidence-Based Intervention REACH Phase 1 | at 12 weeks
  The proportion of eligible patients who enroll in EBI in Phase 1.
Evidence-Based Intervention REACH Phase 2 | at 24 weeks
  The proportion of eligible patients who enroll in EBI in Phase 2.
Participant engagement with dissemination strategies | at 24 weeks
  Proportion of eligible patients who respond to any text message or who talk to a PN
Evidence-Based Intervention Engagement | at 12 weeks from enrollment
  Percent change in the patient's bodyweight, 3 months after enrollment into the Evidence-Based Intervention, among patients who enrolled in the Evidence-Based Intervention.

CONTACTS AND LOCATIONS:
Overall Officials: David Wetter, PhD, Principal Investigator — University of Utah
Locations (1):
- Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schlechter CR, Del Fiol G, Jones DR, Orleans B, Gibson B, Nahum-Shani I, Maxfield E, Locke A, Cornia R, Bradshaw R, Wirth J, Jaggers SJ, Lam CY, Wetter DW. Increasing the reach of evidence-based interventions for weight management and diabetes prevention among Medicaid patients: study protocol for a pilot Sequential Multiple Assignment Randomised Trial. BMJ Open. 2023 Nov 27;13(11):e075157. doi: 10.1136/bmjopen-2023-075157. PMID 38011967